CLINICAL TRIAL: NCT04188080
Title: De-escalation of the Daily Jarlsberg Cheese-dose Related to the Osteocalcin Level in Healthy Women: Estimation of a Maintaining Daily Jarlsberg Cheese-dose
Brief Title: Estimation of a Maintaining Daily Jarlsberg Cheese-dose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meddoc (Other)
Collaborators: Tine (Industry); Norwegian University of Life Sciences (Other)
Responsible Party: Principal Investigator, Prof Stig Larsen, Professor, Meddoc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HV-Jarlsberg/IB
Record Dates: First submitted 2019-12-02; First posted 2019-12-05 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Maintenance Dose; Osteocalcin; Vitamin K Deficiency
Keywords: Jarlsberg cheese
MeSH Terms: conditions — Vitamin K Deficiency

STUDY DESIGN:
Intervention Model Description: Within-patient Response Surface Pathway
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Jarlsberg cheese starting dose (Experimental): The participants obtaining an Osteocalcin increase > 10% during the previous 6 weeks intake of Jarlsberg cheese, will get a percent reduction in the daily cheese-dose equal to the increase in the Osteocalcin level
  Interventions: Dietary Supplement: Jarlsberg Cheese

INTERVENTIONS:
Dietary Supplement: Jarlsberg Cheese — Oral daily intake of Jarlsberg cheese

SUMMARY:
The study objective is to estimate a maintaining daily dose of Jarlsberg cheese in healthy pre-menopausal women obtaining an increase in the osteocalcin level of at least 10% after 6 weeks on maximum efficacy dose (MED) of Jarlsberg cheese.

1.4: Population and sampling The study population consists of Healthy Voluntary (HV) women between 20 years and pre-menopausal age.

The study will be performed as a one-dimensional, within-patient, 3-level Response Surface Pathway (RSP) designed trial with individually adjustment of the dose. Each design period will be 3 weeks. Only HVs obtaining an increase in the osteocalcin level ≥ 10% from baseline after 6 weeks on the MED of 57g Jarlsberg cheese daily will be offered to participate in this de-escalation study.

DETAILED DESCRIPTION:
The recruited HV women fulfilled the inclusion without the exclusion criteria for the study will undergo a screening clinical investigation. The participants will be asked to avoid use of other cheese than the one allocated to in the study, but eat as usual. One week later, the first clinical investigation in the study will take place including blood sampling and measurement of visual signs. The HV women verified to fulfil the criteria for participation and signed the informed consent form will be included in the study. During this first clinical investigation in the study denoted as Day 0, the participants receive a study identification number. The daily intake of cheese will be 57g/day . The trial cheese can be consumed with other food at breakfast, lunch or other meals during the day.

The participants meet for new clinical investigations every third week with measurement of visual signs and blood sampling. The first 12 HVs finalized 6 weeks with daily intake of 57 g Jarlsberg cheese obtaining an increase in the osteocalcin level from baseline ≥10% will be offered participation in this de-escalation study. The results of the osteocalcin analysis after 6 weeks will be ready within one week and the HVs continue on unchanged cheese dose. The HVs participating in this de-escalation study will be included in this part after 7 weeks. The remaining HVs will continue the Jarlsberg cheese intake as prescribed in protocol HV-Jarlsberg/III.

The de-escalation study consists of three design level each of three weeks duration. The analysis of the osteocalcin level taken after three weeks will be ready within one week later. This measurement will be the background for change in the dose for the next design level. During this first week after the three-week period, the HVs will continue on the same cheese dose until the results from the osteocalcin analysis is available.

The HVs included in this de-escalation study will receive a reduced daily dose of Jarlsberg cheese for three weeks in the first design level. The reduction in the daily Jarlsberg cheese dose will be individually calculated. Assume a given HV obtained X % increase in the osteocalcin level during the previous six weeks with a daily dose of 57g. The reduction in the daily Jarlsberg cheese dose for the first design level will be x% [(57*X)/100]. If the osteocalcin level reduces > 10% from the 6-weeks level after 3 weeks on the reduced dose, the dose will be increased for this HV on the second design level. In case the obtained change in the osteocalcin level is ± 10%, the dose will be unchanged. If the osteocalcin level increases > 10 % from the 6-week level, the cheese dose will be reduced for this HV in the second design level. The size of the dose increase or decrease from the first to the second design level depending on the change in the osteocalcin level from the 6-week level and calculated in accordance with the RSP procedure. The change in the osteocalcin level during the second design level will be the basis for calculation of the dose to be used in the third design level. The same procedure as described for the dose-change from the first to the second design level will be used. Clinical investigation and blood sampling will be performed every third week. Osteocalcin and vitamin K will be analysed every third week whereas the haematological and biochemical analysis will be performed at baseline and after 6 and 18 weeks of cheese intake.

The main variable in this study will be osteocalcin measured in serum blood and percent increase in osteocalcin from baseline. Additionally, carboxylated and under carboxylated Osteocalcin and the ratio OR = [Carboxylated / Under Carboxylated] osteocalcin in serum will be central together with the K2 variants MK-7, 8, 9, 9(4H) and vitamin K1. Triglyceride, LDL- and HDL cholesterol, vitamin D and vital signs will be secondary variables. As safety variables, haematological- and biochemical variables and adverse events (AE) will be recorded at each visit.

In accordance with the development of the RSP-procedure, 12 HVs will be included in the study and participate in all the three design levels.

ELIGIBILITY:
Inclusion Criteria:

* Health women (HV) from 20 years of age and pre-menopausal age obtaining an increase in the Osteocalcin Level >10% during 6 weeks daily intake of 57 g Jarlsberg cheese.

Exclusion Criteria:

* Pregnant women
* Known gastrointestinal disorder
* Abnormal liver or kidney function.
* Diabetes
* Suffering from verified cancer
* Under systemic treatment with corticosteroids or other immunosuppressive drugs the last 3 weeks before start of the trial treatment.
* Participating in another clinical trial with pharmaceuticals the last six weeks before start of this trial treatment.
* Lactose intolerance or known milk product allergy
* Not able to understand information.
* Do not want or not able to give written consent to participate in the study.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2020-01-16 (Actual); Primary Completion 2020-06-05 (Actual); Study Completion 2021-07-16 (Actual)

PRIMARY OUTCOMES:
Change in Osteocalcin level | 3 weeks
  Osteocalcin measured as ng/ml in blood serum

SECONDARY OUTCOMES:
Vitamin K | 3 weeks
  Vitamin K measured as ng/ml in blood serum

OTHER OUTCOMES:
Lipid status (Total Cholesterol | 6 weeks
  Total Cholesterol, HDL- and LDL-Cholesterol measured as mmol/L in blood serum

CONTACTS AND LOCATIONS:
Overall Officials: Helge E Lundberg, MD, Principal Investigator — Skjetten Medical Center
Locations (1):
- Skjetten Legesenter, Skjetten, Akershus, Norway

IPD SHARING:
Plan to Share IPD: No